CLINICAL TRIAL: NCT05700604
Title: The Effect of Pancreatic Insufficiency on Hypoglycemia and Glucagon Response in Children With Cystic Fibrosis
Brief Title: Hypoglycemia and Glucagon Response in CF
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Collaborators: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.933
Record Dates: First submitted 2023-01-02; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cystic Fibrosis; Hypoglycemia; Glucagon Deficiency; Pancreatic Insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Hypoglycemia; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis: 10-18 year-old children with Cystic Fibrosis
- Healthy Controls: age and sex matched healthy controls

SUMMARY:
The goal of this clinical trial is to investigate the etiopathogenesis of isolated hypoglycemia and hypoglycemia with abnormal glucose tolerance in children with Cystic Fibrosis (CF) and to evaluate the role of glucagon and pancreatic insufficiency on hypoglycemia in CF. The main questions it aims to answer are:

1. Do isolated hypoglycemia and hypoglycemia with abnormal glucose tolerance have different etiopathogenesis?
2. What is the role of pancreatic insufficiency in these two conditions? Participants were asked to perform 3-h OGTT and to take blood samples. Researchers compared with healthy peers to see if there is isolated hypoglycemia in OGTT and how is the glucagon response to OGTT in healthy peers.

DETAILED DESCRIPTION:
The exact underlying mechanism of hypoglycemia in CF is still unknown. Some recent studies support the delayed and prolonged insulin secretion and impaired counterregulatory hormone response as the reason of reactive hypoglycemia, whereas the others argued an additive effect of an intrinsic factor.

However, the weakness of these limited studies is that nearly all of them included CF patients who had pancreatic insufficiency (PI) and could not reveal the mechanism of hypoglycemia seen in those without PI. In addition, there were no healthy controls for comparison of glucagon secretion in CF patients with hypoglycemia. Moreover, the studies that evaluate the role of glucagon in hypoglycemic CF patients were performed in hypoglycemic adult patients with abnormal glucose tolerance (AGT) and the delayed and prolonged insulin release is expected to be more likely as the reason of hypoglycemia in this setting. Previously, the investigators had demonstrated isolated hypoglycemia in some of the pediatric CF patients during OGTT. In this study, the investigators aimed to further investigate possible mechanisms of hypoglycemia. The investigators hypothesized that the mechanism of isolated hypoglycemia might be different from hypoglycemia seen in patients with AGT. Furthermore, the investigators evaluated the role of pancreatic insufficiency in hypoglycemia of CF patients by analyzing glucose, insulin and glucagon response to a glucose load in CF patients with and without PI.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 year-old children genetically diagnosed with Cystic Fibrosis
* Regularly followed by the department of pediatric endocrinology

Exclusion Criteria:

* Using corticosteroid therapy in the last 3 months
* Those who had acute exacerbation in the last 3 months
* Previously diagnosed with diabetes

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population is the children and adolescents aged 10-18 years with CF who were regularly followed-up at the Pediatric Endocrinology and Diabetes Units.
  The control group was age-matched healthy, diabetes non-diabetic siblings of patients with type 1 diabetes. All the controls were negative for β-cell autoantibodies (anti-glutamic acid decarboxylase, islet cell antibody, and insulin antibody).
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change of glucose level | 0-30-60-90-120-150-180.minutes of oral glucose loading
  A 3 hour Oral Glucose Tolerance Test (OGTT) was used to evaluate changing and it was performed in the morning following overnight fasting of ≥8 hours. All participants (CF patients and controls) received oral glucose solution (1.75 g/kg; max: 75 g) in 10 minutes.
Change of insulin level | 0-30-60-90-120-150-180.minutes of oral glucose loading
  A 3 hour Oral Glucose Tolerance Test (OGTT) was used to evaluate changing and it was performed in the morning following overnight fasting of ≥8 hours. All participants (CF patients and controls) received oral glucose solution (1.75 g/kg; max: 75 g) in 10 minutes.
Change of glucagon level | 0-60-120-150-180.minutes of oral glucose loading
  A 3 hour Oral Glucose Tolerance Test (OGTT) was used to evaluate changing and it was performed in the morning following overnight fasting of ≥8 hours. All participants (CF patients and controls) received oral glucose solution (1.75 g/kg; max: 75 g) in 10 minutes.

SECONDARY OUTCOMES:
HbA1c | 0.minute of oral glucose loading
  It was measured by high-performance liquid chromatographic (HPLC) method from venous blood sample
C-reactive protein (CRP) | 0.minute of oral glucose loading
  It was measured by ELISA from venous blood sample
Cortisol | 0-180.minutes of oral glucose loading
  The response to hypoglycemia was evaluated during 3 hour Oral Glucose Tolerance Test (OGTT)
Forced expiratory volume in 1 second (FEV1) | Within 2 weeks before OGTT
  It was measured by spirometry
Body Mass Index (BMI) | Within 24 hours of OGTT
  It was calculated as weight (kg)/height (m)2

CONTACTS AND LOCATIONS:
Overall Officials: Belma Haliloglu, MD,PhD, Study Director — Marmara University, School of Medicine, Department of Pediatric Endocrinology
Locations (1):
- Marmara University, School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All data except the participants' name-surname can be shared with the other researchers

REFERENCES:
- [Result] Kilberg MJ, Sheikh S, Stefanovski D, Kubrak C, De Leon DD, Hadjiliadis D, Rubenstein RC, Rickels MR, Kelly A. Dysregulated insulin in pancreatic insufficient cystic fibrosis with post-prandial hypoglycemia. J Cyst Fibros. 2020 Mar;19(2):310-315. doi: 10.1016/j.jcf.2019.07.006. Epub 2019 Aug 8. PMID 31402215
- [Result] Kilberg MJ, Harris C, Sheikh S, Stefanovski D, Cuchel M, Kubrak C, Hadjiliadis D, Rubenstein RC, Rickels MR, Kelly A. Hypoglycemia and Islet Dysfunction Following Oral Glucose Tolerance Testing in Pancreatic-Insufficient Cystic Fibrosis. J Clin Endocrinol Metab. 2020 Oct 1;105(10):3179-89. doi: 10.1210/clinem/dgaa448. PMID 32668452
- [Result] Aitken ML, Szkudlinska MA, Boyko EJ, Ng D, Utzschneider KM, Kahn SE. Impaired counterregulatory responses to hypoglycaemia following oral glucose in adults with cystic fibrosis. Diabetologia. 2020 May;63(5):1055-1065. doi: 10.1007/s00125-020-05096-6. Epub 2020 Jan 29. PMID 31993716
- [Result] Armaghanian N, Hetherington J, Parameswaran V, Chua EL, Markovic TP, Brand-Miller J, Steinbeck K. Hypoglycemia in cystic fibrosis during an extended oral glucose tolerance test. Pediatr Pulmonol. 2020 Dec;55(12):3391-3399. doi: 10.1002/ppul.25081. Epub 2020 Oct 16. PMID 32955169

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT05700604/Prot_SAP_ICF_000.pdf